CLINICAL TRIAL: NCT05131945
Title: GRAvity- Versus Wall Suction-drIven Large Volume Thoracentesis: a RAndomized Controlled Study (GRAWITAS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2018-0654; NCI-2021-13202 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-10-27; First posted 2021-11-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thoracentesis; Pleural Effusions, Chronic; Pulmonary Edema
MeSH Terms: conditions — Pleural Effusion; Bronchiolitis Obliterans Syndrome; Pulmonary Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Standard Suction Thoracentesis (Experimental): treatment techniques suction is a standard of care and used for draining fluid around the lung.
  Interventions: Other: Standard Suction Thoracentesis; Other: Gravity Thoracentesis
- Group 2: Gravity Thoracentesis. (Experimental): treatment techniques (gravity ) is a standard of care and used for draining fluid around the lung.
  Interventions: Other: Standard Suction Thoracentesis; Other: Gravity Thoracentesis

INTERVENTIONS:
Other: Standard Suction Thoracentesis — a procedure that removes excess fluid from the space in between your lungs and chest wall
Other: Gravity Thoracentesis — a procedure that removes excess fluid from the space in between your lungs and chest wall

SUMMARY:
The primary objective of this study is to compare gravity-driven versus wall suction-driven large volume therapeutic thoracentesis on the development of chest discomfort during the procedure.

This study is a multicenter, single-blinded, randomized controlled trial designed to compare chest discomfort between gravity-driven and wall suction-driven therapeutic thoracentesis. Patients will be stratified by study centers, and randomly assigned to intervention and control arms; and will remain blinding to their group assignment during the procedure.

DETAILED DESCRIPTION:
Aims and Objectives:

The primary objective of this study is to compare gravity-driven versus wall suction-driven large volume therapeutic thoracentesis on the development of chest discomfort during the procedure.

Expected Outcomes:

We anticipate that gravity driven therapeutic thoracentesis will result in improved clinical outcomes compared to wall suction driven thoracentesis, defined by less chest discomfort throughout the procedure as measured at 5 minutes post-procedure (primary endpoint).

Primary endpoint:

The Global Pain Score will be determined at 5 minutes post-procedure using a VAS 0-100 and represents the pain experienced by the patient during the entire procedure from the beginning to the 5-minute post-procedure assessment ("On average, how much discomfort have you felt during the procedure?"). The primary endpoint is defined as the overall procedural chest pain scored 5 minutes following the procedure.

This study is a randomized controlled trial designed to compare the changes of chest pain scores between gravity-driven therapeutic thoracentesis and wall suction-driven thoracentesis. The estimated minimal clinically important difference of the change is 10.

Secondary endpoints:

1. Duration of procedure timed from the beginning of fluid drainage to catheter removal.
2. Differences in narcotics used after the procedure.
3. Incidence of pneumothorax detected on the post procedural CXR
4. Incidence of clinically apparent re-expansion pulmonary edema
5. Incidence of radiographically apparent re-expansion pulmonary edema detected on the post procedural CXR

ELIGIBILITY:
Inclusion criteria:

1. Referral to pulmonary services for large-volume thoracentesis
2. Presence of a symptomatic moderate or large free-flowing (non-septated) pleural effusion on the basis of:

   1. Chest radiograph: effusion filling ≥ 1/3 the hemithorax, OR
   2. CT-scan: maximum AP depth of the effusion ≥ 1/3 of the AP dimension on the axial image superior to the hemidiaphragm, including atelectatic lung completely surrounded by effusion, OR Ultrasound: effusion spanning at least three interspaces, with depth of 3 cm or greater in at least one intercostal space, while the patient sits upright.
3. Age >/= 18

Exclusion criteria:

1. Inability to provide informed consent
2. Study subject has any disease or condition that interferes with safe completion of the study including:

   1. Coagulopathy, with criteria left at the discretion of the operator
   2. Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the attending physicians
3. Pleural effusion is smaller than expected on bedside pre-procedure ultrasound
4. Referral is for diagnostic thoracentesis only
5. Presence of more than minimal septations and/or loculations( more than 3) on bedside pre-procedure ultrasound
6. Inability to sit for the procedure
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
The overall procedural chest pain questionnaire | through study completion, an average of 1 year
  The Global Pain Score will be determined at 5 minutes post-procedure using a VAS 0-100 and represents the pain experienced by the patient during the entire procedure from the beginning to the 5-minute post-procedure assessment

CONTACTS AND LOCATIONS:
Overall Officials: Horianna Grosu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shojaee S, Pannu J, Yarmus L, Fantin A, MacRosty C, Bassett R Jr, Debiane L, DePew ZS, Faiz SA, Jimenez CA, Avasarala SK, Vakil E, DeMaio A, Bashoura L, Keshava K, Ferguson T, Adachi R, Eapen GA, Ost DE, Bashour S, Khan A, Shannon V, Sheshadri A, Casal RF, Evans SE, Pew K, Castaldo N, Balachandran DD, Patruno V, Lentz R, Pai C, Maldonado F, Roller L, Ma J, Zaveri J, Los J, Vaquero L, Ordonez E, Yermakhanova G, Akulian J, Burks C, Almario RR, Sauve M, Pettee J, Noor LZ, Arain MH, Grosu HB. Gravity- vs Wall Suction-Driven Large-Volume Thoracentesis: A Randomized Controlled Study. Chest. 2024 Dec;166(6):1573-1582. doi: 10.1016/j.chest.2024.05.046. Epub 2024 Jul 18. PMID 39029784
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org